CLINICAL TRIAL: NCT00959634
Title: Pharmacokinetic Study of ABT-126 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Robert Lenz, MD, PhD / Project Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M11-988
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Dose 1 BID
  Interventions: Drug: ABT-126
- 2 (Experimental): Dose 2 BID
  Interventions: Drug: ABT-126
- 3 (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-126 — Dose administered twice daily on Study Days 1-10
  Arms: 1; 2
Drug: Placebo — Dose administered twice daily on Study Days 1-10
  Arms: 3

SUMMARY:
This is a study to investigate the process by which ABT-126 is absorbed, distributed, metabolized and eliminated by the body of a healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 50 years of age
* If female, subject must be postmenopausal for at least 2 years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* If male, subject must be surgically sterile (vasectomy) or agrees to use a barrier method (i.e., condom) of birth control starting on the first day of confinement until 30 days after the last study drug administration

Exclusion Criteria:

* Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements on a regular basis
* History of diabetes, cancer (except basal cell carcinoma of the skin), or any clinically significant cardiovascular, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, neurologic or psychiatric disease or disorder
* Presence of any uncontrolled medical illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (e.g., clinical laboratory tests, vital signs, adverse events assessment, physical examination, brief neurological examination) | One day before dosing through day of last dose and up to 6 days after last dose
ABT-126 levels in blood (plasma) | First dose through last dose and up to 192 hours after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 22863, Austin, Texas, United States